CLINICAL TRIAL: NCT00608504
Title: Biobehavioral Study of Opioid Drug Seeking Behavior: Study 3
Brief Title: Effects of Environmental Factors on Opiate Drug Choice in Opioid Dependent Individuals.
Acronym: DSC
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Principal Investigator, Wayne State University
Other Study IDs: NIDA-15462-3; R01DA015462-03 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Behavioral Economics; Drug self administration; Opioid
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose is to study how certain factors, including money, the amount of drug available and the amount of work effort, affect opiate drug choice.

DETAILED DESCRIPTION:
A drug dependent person chooses to take drug more often (and suffer its long-term bad consequences) than choosing to engage in healthy activities (which have better long-term consequences). The present research will be conducted in a controlled laboratory setting with heroin abusers who are not seeking treatment to understand what factors guide their choices.

This research focuses on environmental (i.e. non-medication) factors that affect choosing a drug versus money. Findings from this research are likely to be important in developing a theoretical and practical basis for behavioral interventions as part of drug abuse treatment. HYD is a drug that is currently used as a cough suppressant and to relieve pain.

Participants in this observational study will take part in multiple trials in which they have the opportunity to choose HYD or money. On the first two experimental days, prior to choice sessions, participants will receive a sample of the drug doses that can be chosen. During test sessions, participants will have 12 opportunities to choose either drug or money. Participants will use a computer to earn choices. Respiration rate, oxygen saturation, heart rate, and blood pressure will be monitored throughout choice trials. Self-report questionnaires will be completed at different times during the study.

Participants will be maintained on buprenorphine throughout the study, with a minimum 2-week lead before the experiment, and a fixed 3-week detoxification after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependent, as determined by structured clinical interview for DSM-IV (SCID) and Addiction Severity Index (ASI)
* Positive urine test for opiates
* Willing to use an adequate form of contraception for the duration of the study.
* Reads and writes English

Exclusion Criteria:

* Psychiatric illness, as determined by the DSM-IV criteria
* History of or current neurological disease, including structural abnormalities, seizures, infection, peripheral neuropathy, and head traumas
* History of cardiovascular disease, myocardial infarction, chest pain, or edema
* Systolic blood pressure greater than 160mm HG or less than 95 mm HG: PR diastolic blood pressure greater than 95 mm HG.
* Pulmonary disease, including obstructive pulmonary disease, Cor pulmonale, tuberculosis, and asthma
* Systemic disease (e.g. endocrinopathies, liver or kidney failure, myxedema, hypothyroidism, Addison's disease, autoimmune disease)
* Current alcohol or sedative drug dependence
* Pregnant or breast feeding
* Currently receiving treatment for opioid dependence
* Known phobia of injections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Heroin dependent research volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Woodcock EA, Lundahl LH, Burmeister M, Greenwald MK. Functional mu opioid receptor polymorphism (OPRM1 A(118) G) associated with heroin use outcomes in Caucasian males: A pilot study. Am J Addict. 2015 Jun;24(4):329-35. doi: 10.1111/ajad.12187. Epub 2015 Apr 24. PMID 25911999
- [Derived] Stoltman JJ, Woodcock EA, Lister JJ, Greenwald MK, Lundahl LH. Exploration of the telescoping effect among not-in-treatment, intensive heroin-using research volunteers. Drug Alcohol Depend. 2015 Mar 1;148:217-20. doi: 10.1016/j.drugalcdep.2015.01.010. Epub 2015 Jan 19. PMID 25630964
- [Derived] Greenwald MK, Steinmiller CL, Sliwerska E, Lundahl L, Burmeister M. BDNF Val(66)Met genotype is associated with drug-seeking phenotypes in heroin-dependent individuals: a pilot study. Addict Biol. 2013 Sep;18(5):836-45. doi: 10.1111/j.1369-1600.2011.00431.x. Epub 2012 Feb 16. PMID 22339949